CLINICAL TRIAL: NCT00848861
Title: A Trial Comparing Propofol to Midazolam Plus Meperidine Sedation for Outpatient Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Dina Kao, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2-kao
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Sedation
Keywords: propofol sedation; colonoscopy; recovery time; recovery time after sedation for colonoscopy
MeSH Terms: interventions — Propofol; Midazolam; Meperidine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 propofol (Active Comparator)
  Interventions: Drug: propofol (sedation for outpatient colonoscopy)
- 2 midazolam plus meperidine (Active Comparator)
  Interventions: Drug: midazolam plus meperidine (sedation for outpatient colonoscopy)

INTERVENTIONS:
Drug: propofol (sedation for outpatient colonoscopy)
  Arms: 1 propofol
Drug: midazolam plus meperidine (sedation for outpatient colonoscopy)
  Arms: 2 midazolam plus meperidine

SUMMARY:
-to determine if propofol sedation leads to shorter recovery times compared to traditional sedation using midazolam plus meperidine

DETAILED DESCRIPTION:
Colonoscopy is an important diagnostic and therapeutic procedure. It is an invasive procedure, not well tolerated by most patients if performed without sedation. There is considerable variability in the practice of sedation for endoscopic procedures worldwide. There are some centers which perform a significant proportion of gastroscopies and colonoscopies without sedation. On the other hand, general anesthesia is given to more than 90% of patients undergoing colonoscopy in France. Most centers do use conscious sedation, usually in the form of benzodiazepines and/or narcotics, with propofol sedation reserved for difficult cases. Benzodiazepines and narcotics are effective and safe. However, the onset of sedation can be delayed, and in some patients conscious sedation is inadequate, resulting in a poor experience with the procedure. Moreover, there are significant post-sedation side effects, such as nausea, vomiting, and prolonged recovery period. This can substantially increase procedure costs due to the need for prolonged monitoring after endoscopy.

Propofol, a general anesthetic agent, has been routinely used in various procedures and surgeries. It has a fast onset of action (within 30-60 seconds), a short half life (1.8-4.1 minutes) but a narrow therapeutic window. The current package insert of propofol states that only persons trained in the administration of general anesthesia should administer propofol and these physicians should not be involved in the procedure so that patients can be continuously and properly monitored due to the risk of respiratory depression. No deaths associated with propofol sedation have been reported since it was first introduced in gastrointestinal endoscopy in the mid 1980. However, need for mechanical ventilation as a result of propofol sedation has been reported. In a number of small trials propofol was shown to have a superior recovery profile following various endoscopic procedures including gastroscopy, colonoscopy and endoscopic retrograde cholangiopancreatography (ERCP). Indeed, propofol sedation is now used routinely in elective adult procedures in some centers. However, the lower cost of recovery is offset by the need for an anesthesiologist. Therefore, the use of propofol sedation is limited to selected endoscopic procedures or patients.

Although a number of small randomized trials have explored the efficacy of propofol sedation, the evidence is not definitive. Thus we conducted this study to determine if propofol sedation leads to shorter recovery times in elective outpatient colonoscopy compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* outpatient colonoscopy

Exclusion Criteria:

* allergy to propofol , midazolam, meperidine, eggs or soybean
* history of colonic resection
* inability to understand spoken/written English
* dementia
* pregnancy
* unwillingness to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2006-02; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
recovery time

SECONDARY OUTCOMES:
procedure time
patient satisfaction
adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Dina Kao, MD, Principal Investigator — University of Alberta; Eoin Lalor, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Vijan S, Inadomi J, Hayward RA, Hofer TP, Fendrick AM. Projections of demand and capacity for colonoscopy related to increasing rates of colorectal cancer screening in the United States. Aliment Pharmacol Ther. 2004 Sep 1;20(5):507-15. doi: 10.1111/j.1365-2036.2004.01960.x. PMID 15339322
- [Background] Trummel J. Sedation for gastrointestinal endoscopy: the changing landscape. Curr Opin Anaesthesiol. 2007 Aug;20(4):359-64. doi: 10.1097/ACO.0b013e32827ab467. PMID 17620846
- [Background] Riphaus A, Stergiou N, Wehrmann T. Sedation with propofol for routine ERCP in high-risk octogenarians: a randomized, controlled study. Am J Gastroenterol. 2005 Sep;100(9):1957-63. doi: 10.1111/j.1572-0241.2005.41672.x. PMID 16128939
- [Background] Vargo JJ, Zuccaro G Jr, Dumot JA, Shermock KM, Morrow JB, Conwell DL, Trolli PA, Maurer WG. Gastroenterologist-administered propofol versus meperidine and midazolam for advanced upper endoscopy: a prospective, randomized trial. Gastroenterology. 2002 Jul;123(1):8-16. doi: 10.1053/gast.2002.34232. PMID 12105827
- [Background] Kulling D, Fantin AC, Biro P, Bauerfeind P, Fried M. Safer colonoscopy with patient-controlled analgesia and sedation with propofol and alfentanil. Gastrointest Endosc. 2001 Jul;54(1):1-7. doi: 10.1067/mge.2001.116174. PMID 11427833
- [Background] Lee DW, Chan AC, Sze TS, Ko CW, Poon CM, Chan KC, Sin KS, Chung SC. Patient-controlled sedation versus intravenous sedation for colonoscopy in elderly patients: a prospective randomized controlled trial. Gastrointest Endosc. 2002 Nov;56(5):629-32. doi: 10.1067/mge.2002.128919. PMID 12397267
- [Background] Moerman AT, Foubert LA, Herregods LL, Struys MM, De Wolf DJ, De Looze DA, De Vos MM, Mortier EP. Propofol versus remifentanil for monitored anaesthesia care during colonoscopy. Eur J Anaesthesiol. 2003 Jun;20(6):461-6. doi: 10.1017/s0265021503000723. PMID 12803263